CLINICAL TRIAL: NCT02471339
Title: Acceptance and Commitment Training for Adolescents and Young Adults With Neurofibromatosis Type 1, Plexiform Neurofibromas, and Chronic Pain: A Phase III Clinical Trial
Brief Title: Acceptance and Commitment Training for Adolescents and Young Adults With Neurofibromatosis Type 1, Plexiform Neurofibromas, and Chronic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Staci Peron, Ph.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 150142; 15-C-0142
Record Dates: First submitted 2015-06-12; First posted 2015-06-15 (Estimated); Results first posted 2021-12-06 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-05

CONDITIONS: Neurofibromatosis Type 1; Plexiform Neurofibromas
Keywords: Psychological Intervention; Coping; Mindfulness; Randomized
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma, Plexiform | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1/Acceptance and Commitment Therapy (ACT) Group (Experimental): 2 Acceptance and Commitment Therapy (ACT) Training Sessions followed by weekly emails and video chats.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT)
- 2/Waitlist (WL) Group (Active Comparator): Waitlist group - no intervention for first 8 weeks (then will receive Acceptance and Commitment Therapy (ACT) intervention as Arm 1)
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT)

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) — Acceptance and Commitment Therapy (ACT), a newer generation of cognitive-behavioral therapy, focuses on encouraging individuals to engage in more adaptive ways of coping with pain.

SUMMARY:
Background:

- People with neurofibromatosis type I (NF1) and plexiform neurofibroma (PN) tumors often have chronic pain that his hard to control. People usually take medicines for the pain, but they may not work well and might cause side effects. A new strategy called Acceptance and Commitment Training (ACT) may help these people cope with chronic pain. ACT focuses on things like values and living in the moment.

Objective:

- To see if Acceptance and Commitment Training improves pain coping in people with NF1 pain.

Eligibility:

- People age 16-34 who have NF1, 1 or more PN tumors, and pain that interferes with their daily functioning.

Design:

* Participants will be screened with a physical exam, medical history, and questions about their pain.
* Participants will fill out questionnaires about their pain and feelings. Their heart rate will be measured via electrocardiogram (ECG).
* Participants will be divided into 2 groups randomly. One will wait 8 weeks.
* The other will start training right away.
* Participants will have 2 two-hour sessions with an ACT trainer. They will learn techniques for setting goals based on personal values and other ways to cope with pain. They will get a workbook and a compact disc (CD) to take home for practice.
* Participants will do practice exercises at home between sessions. They will get weekly emails with a practice exercise. They will join video chat sessions via home computer with their trainer.
* All participants will return to National Institutes of Health (NIH) after 8 weeks for questionnaires and an ECG. The wait group will then start training. They will return 8 weeks later for questionnaires and an ECG.
* Six months later, they will complete questionnaires from home by computer.

DETAILED DESCRIPTION:
BACKGROUND:

* Neurofibromatosis type 1 (NF1) is a genetic disorder that affects approximately 1 in 3,500 individuals.
* A number of common clinical manifestations, including plexiform neurofibromas, can cause frequent and significant pain and impact quality of life.
* Often, NF1-related pain is not well-controlled with medication and many of the medications cause significant side effects.
* To our knowledge, only one prior study (by our group) has examined the effectiveness of a psychological intervention for chronic pain in adolescents and young adults (AYA) with NF1.
* Acceptance and Commitment Therapy (ACT), a newer generation of cognitive-behavioral therapy, focuses on encouraging individuals to engage in more adaptive ways of coping with pain.
* The goal of ACT is not to eliminate the person's pain, but to optimize the person's functioning despite their pain

OBJECTIVES:

-To compare pain interference mean score changes from baseline to 8 weeks between the ACT intervention group and the waitlist (WL) group.

ELIGIBILITY:

* Patients 16 - 59 years of age with a confirmed diagnosis of NF1 and greater than or equal to 1 plexiform neurofibroma (PN).
* The patient must obtain a mean score of 2.0 or higher or a score of 3 on three or more items on the Pain Interference Index, and report having pain that interferes with functioning for at least three months.
* The patient must have regular access to a computer or tablet with internet access.

DESIGN:

* This is a psychological intervention study to determine the potential benefit of ACT on pain interference, with patients randomized to the ACT intervention or a wait-list control group.
* Patients will come to the National Institutes of Health (NIH) for a 2-day visit (Time 1). After baseline assessments (questionnaires and ECG) are completed, participants in the ACT group will take part in two 2-hour ACT training sessions. At home, this group will receive weekly emails through week 8, and will participate in further ACT training/educational sessions via video chat at weeks 2, 4, and 6.
* All patients will return to the NIH at week 8 (Time 2) to complete follow-up questionnaires and ECG. At this time, the WL group will cross over and receive the ACT intervention (in-person sessions, weekly emails, and video chat sessions). All patients will complete questionnaires again from home six months following the completion of the intervention.
* To detect a change of .68 standard deviation on the primary outcome measure between the two groups at .80 power, 41 patients per group are needed.

ELIGIBILITY:
* INCLUSION CRITERIA FOR PARTICIPANT

  1. Patients must be between 16 and 59 years of age at the time of the baseline assessment. Because the research on the effectiveness of Acceptance and Commitment Therapy (ACT) with younger children is still emerging, children 15 and younger will be excluded from the present study.
  2. Diagnosis of Neurofibromatosis Type 1 (NF1) through germline mutation OR clinical diagnosis; for the clinical diagnosis of NF1 all study subjects must have two or more diagnostic criteria for NF1 listed below (National Institutes of Health (NIH) Consensus Conference):

     * Six or more cafe-au-lait spots (greater than or equal to 0.5 cm in prepubertal subjects or greater than or equal to 1.5 cm in postpubertal subjects)
     * Greater than or equal to 2 neurofibromas or 1 plexiform neurofibroma
     * Freckling in the axilla or groin
     * Optic glioma
     * Two or more Lisch nodules
     * A distinctive bony lesion (dysplasia of the sphenoid bone or dysplasia or thinning of long bone cortex)
     * A first-degree relative with NF1
  3. Participants must have documentation of a plexiform neurofibromas (PN), based on either clinical exam or imaging.
  4. Patient must self-report having chronic pain for at least the past 3 months that has interfered with their daily functioning, as assessed by the Pain Interference Index (must get a mean score of 2.0 or higher, or score a 3 on three or more individual items).
  5. Patients must have regular access to a computer or tablet with internet access.
  6. Ability of subject or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document.
  7. No anticipated major changes in their pain treatment regimen (i.e., new class of pain medication starting or change in the class of pain medication) or enrollment on a new treatment study presumed to impact pain in the near future.
  8. Subjects must be able to read and comprehend the English language, since the highly trained ACT therapists are not fluent enough to conduct the trainings in Spanish or other languages.

EXCLUSION CRITERIA FOR PARTICIPANT

1. In the opinion of the Principal Investigator (PI) or an Associate Investigator (AI), the subject has significant cognitive or emotional difficulties that would prevent them from being able to understand and/or participate fully in the intervention or the measures.
2. Subjects who are participating in any other treatment studies, either medical or behavioral, specifically for pain management.
3. Subjects who began a medical intervention for treatment of their disease that has a possible impact on pain (including Mitogen-activated Protein/Extracellular Signal-regulated Kinase Kinase (MEK) trials) will not be eligible until after one year on the medical treatment; at that time, eligibility will be discussed with the PI of the medical study to assess the stability of the patient s pain and whether further pain-related changes due to the medical treatment are likely.
4. Inability to travel to the NIH, for example, due to physical limitations, for the in-person evaluation(s).

No groups in regards to gender, race, or ethnicity are being excluded from participation in the trial.

Ages: 16 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2015-07-07 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2020-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Staci M Peron, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The authors will make the data, protocol, and statistical plan available upon request. Also share raw data per researchers request to access the IPD via the online platform Yale University Open Data Access (YODA).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The protocol, SAP, and data will be shared when published on clinicaltrials.gov indefinitely.
Access Criteria: http://yoda.yale.edu/

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-C-0142.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 66/67 are enrolled on this study because one participant was deemed ineligible and taken off study.
Period: Overall Study
Arm/Group | 1/Acceptance and Commitment Therapy (ACT) Group | 2/Waitlist (WL) Group
Started | 32 | 34
Completed | 30 | 34
Not Completed | 2 | 0
Not completed — Did not provide follow-up data | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1/Acceptance and Commitment Therapy (ACT) Group | 2/Waitlist (WL) Group | Total
Number analyzed (Participants) | 32 | 34 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 3 | 6
  Between 18 and 65 years | 29 | 31 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.09 (11.74) | 28.88 (10.35) | 29.98 (11.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 17 | 40
  Male | 9 | 17 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 28 | 29 | 57
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 6 | 9
  White | 23 | 22 | 45
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 32 | 34 | 66

OUTCOME MEASURES:

1. Primary Outcome: Mean Pain Interference Mean Score Change From Baseline to 8 Weeks Between the Acceptance and Commitment Therapy Intervention Group and the Waitlist Group
Description: Pain interference mean score changes were compared between the two groups from baseline to 8 weeks using the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Scale.T-scores typically can range from 0 to 100, with "average" scores ranging from 41-59. No subscales are included in this measure. Higher scores indicate more pain interference (worse).
  A two-way repeated-measures analysis of covariance (ANCOVA) was used to examine changes between groups from baseline to the 8-week follow-up.
Time Frame: Baseline and 8 weeks
Population: 30/34 were analyzed in the Waitlist group because 2 participants were withdrawn from final analyses due to medical contraindications identified immediately after the post-intervention follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1/Acceptance and Commitment Therapy (ACT) Group | 2/Waitlist (WL) Group
Number analyzed (Participants) | 32 | 30
score on a scale
  Baseline | 61.93 (5.9) | 62.87 (5.9)
  8 weeks | 56.89 (6.4) | 61.21 (6.7)
Statistical Analysis 1: Comparison: 1/Acceptance and Commitment Therapy (ACT) Group vs 2/Waitlist (WL) Group; Analysis of covariance. Analyses for primary and secondary outcomes were two-tailed and alpha was set to 0.05. An a priori analysis suggested that, to detect a change of .68 standard deviation on the primary outcome measure between the two groups at .80 power, 41 patients per group would be needed; Test type: Superiority; p = 0.05, ANCOVA

2. Secondary Outcome: Change in Quality of Life (QOL) for Physical Functioning
Description: Baseline to post-treatment changes in disease-related quality of life was assessed various aspects of quality of life using a subscale from the Pediatric Quality of Life Inventory (PedsQL) Neurofibromatosis Type 1 (NF) Module adult questionnaire which uses a 0-4 Likert scale (0= never, 4 = almost always). Physical Functioning (7 items; possible range 0-28) subscale was administered. Higher scores are worse. Mean scores are linearly transformed to a 0-100 scale, and then were compared to means and standard deviations of a normative group of patients with Neurofibromatosis Type 1.
Time Frame: Baseline and 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1/Acceptance and Commitment Therapy (ACT) Group | 2/Waitlist (WL) Group
Number analyzed (Participants) | 32 | 30
score on a scale
  Baseline | 37.97 (19.4) | 38.17 (21.9)
  8 weeks | 42.39 (21.9) | 47.70 (25.5)
Statistical Analysis 1: Comparison: 1/Acceptance and Commitment Therapy (ACT) Group vs 2/Waitlist (WL) Group; Test type: Superiority; p = 0.05, ANCOVA

3. Secondary Outcome: Mean Pain Acceptance Pre- and Post-treatment
Description: Measure of Pain Acceptance pre- and post-treatment was assessed by the Chronic Pain Acceptance Questionnaire (CPAQ) to determine if participants can accept his or her pain. Participants answer 20 questions on a 0 (never true) to 6 (always true) rating scale, with higher scores indicating higher levels of acceptance. Scores are obtained on two subscales (Activities Engagement and Pain Willingness) and an Acceptance Total scale. Only the total score was analyzed for this study. Scores can range from 0 to 120, with higher scores indicating more acceptance (better).
Time Frame: Baseline and 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1/Acceptance and Commitment Therapy (ACT) Group | 2/Waitlist (WL) Group
Number analyzed (Participants) | 32 | 30
score on a scale
  Baseline | 58.78 (14.9) | 55.60 (14.8)
  8 Weeks | 71.91 (15.7) | 58.07 (15.9)

4. Secondary Outcome: Change in Disease-related Pain Severity and Overall Tumor Pain
Description: Pre and post changes in disease-related pain severity and overall tumor pain was assessed using the Numeric Rating Scale - 11 (NRS-11). Two questions rate pain severity on a scale of 0 (no pain) to 10 (worst pain imaginable). For both questions, higher scores = more pain. The two questions are examined separately, there is no total score across items.
Time Frame: Baseline and 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1/Acceptance and Commitment Therapy (ACT) Group | 2/Waitlist (WL) Group
Number analyzed (Participants) | 32 | 30
score on a scale
  Baseline disease-related pain severity | 7.52 (1.8) | 7.39 (1.6)
  8 weeks disease-related pain severity | 6.8 (2.6) | 6.97 (2.5)
  Baseline overall tumor pain | 7.53 (1.76) | 7.03 (2.58)
  8 weeks overall tumor pain | 6.81 (2.56) | 5.87 (2.62)

5. Secondary Outcome: Change in Quality of Life (QOL) for Daily Activities
Description: Baseline to post-treatment changes in disease-related quality of life, including Daily Activities was assessed using a subscale from the Pediatric Quality of Life Inventory (PedsQL) Neurofibromatosis Type 1 (NF) Module adult questionnaire which uses a 0-4 Likert scale (0= never, 4 = almost always). Daily Activities (12 items; possible range 0-48) subscale was administered. Higher scores are worse. Mean scores are linearly transformed to a 0-100 scale, and then were compared to means and standard deviations of a normative group of patients with Neurofibromatosis Type 1.
Time Frame: Baseline and 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1/Acceptance and Commitment Therapy (ACT) Group | 2/Waitlist (WL) Group
Number analyzed (Participants) | 32 | 30
score on a scale
  Baseline | 84.3 (13.6) | 80.5 (14.7)
  8 weeks | 87.2 (12.8) | 80.4 (20.2)
Statistical Analysis 1: Comparison: 1/Acceptance and Commitment Therapy (ACT) Group; Test type: Superiority; p = .05, t-test

6. Secondary Outcome: Change in Disease-related Depression
Description: Pre and post changes in disease-related depression was assessed using the 20-item Center for Epidemiological Studies - Depression scale (CES-D). Participants rate symptoms they have experienced in the past week and items are scored on a 0 (rare or none of the time) to 3 (most of all of the time) scale. Individual responses yield scores on four subscales: depressive affect, positive affect, somatic activity, and interpersonal. A total depression score is obtained that can range from 0 to 60, with higher scores representing worse depressive symptoms.
Time Frame: Baseline and 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1/Acceptance and Commitment Therapy (ACT) Group | 2/Waitlist (WL) Group
Number analyzed (Participants) | 32 | 30
score on a scale
  Baseline | 21.88 (12.3) | 25.40 (12.5)
  8 weeks | 18.47 (10.5) | 22.53 (11.9)

7. Secondary Outcome: Change in Pain-related Anxiety
Description: Pre and post changes in disease-related pain-related anxiety was assessed by the Pain Anxiety Assessment Scale - 20 (PASS-20). Items are answered on a 6-point Likert scale with anchors of "never" and "always" which provides a total score and scores on four subscales for Cognitive Anxiety, Pain-related Fear, Escape and Avoidance, and Physiological Anxiety. We only examined the total score on this measure, which can range from 0 to 100; higher scores indicate more anxiety.
Time Frame: Baseline and 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1/Acceptance and Commitment Therapy (ACT) Group | 2/Waitlist (WL) Group
Number analyzed (Participants) | 32 | 30
score on a scale
  Baseline | 52.44 (20.6) | 52.57 (21.5)
  8 weeks | 42.4 (22.3) | 45.37 (20.7)

8. Secondary Outcome: Change in Heart Rate Variability (HRV)
Description: Pre and post changes in disease-related HRV was assessed using an electrocardiogram (EKG). An EKG records electrical signals from your heart. The EKG reading will occur for 5 minutes while the patient is lying down and measurements, including the standard deviation of the average NN (normal-to-normal) interval (SDANN) and the square root of the mean squared differences of successive NN intervals is recorded, resulting in a metric of parasympathetically mediated (high frequency) HRV in milliseconds.
Time Frame: Baseline and 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | 1/Acceptance and Commitment Therapy (ACT) Group | 2/Waitlist (WL) Group
Number analyzed (Participants) | 32 | 30
milliseconds
  Baseline | 68.63 (64.8) | 94.74 (119.4)
  8 weeks | 88.11 (88.0) | 82.00 (99.8)

9. Secondary Outcome: Pain Interference Patient-Reported Outcomes Measurement Information System (PROMIS) II
Description: The psychometric properties of the pain interference measure PROMIS was administered to assess pain interference. And adult (18-59 years) and pediatric (16 -17 years) questionnaire was administered to assess how pain interferes with sleep, mood, and leisure activities for instance. Items were formatted on 0-4 Likert scales (0 = Never, 4 = Almost Always) and transformed to T-scores. The PROMIS Pain Interference Scale takes less than 5 minutes to complete and is required of all participants. T-scores typically range from the 20s to 80s with a mean of 50 and standard deviation of 10 ("average" scores range from 40 - 60). No subscales are included in this measure. Higher scores indicate more pain interference (worse). The pediatric and adult versions are made to be parallel so we analyzed all participants together across ages. A two-way repeated-measures analysis of variance (ANOVA) was used to examine changes between groups from baseline to the 8-week follow-up.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | 1/Acceptance and Commitment Therapy (ACT) Group | 2/Waitlist (WL) Group
Number analyzed (Participants) | 32 | 30
T-scores
  Adult & Pediatric - Baseline | 61.9 (4.9) | 62.9 (5.9)
  Adult & Pediatric - 8 weeks | 56.9 (6.4) | 61.2 (6.9)
Statistical Analysis 1: Comparison: 1/Acceptance and Commitment Therapy (ACT) Group vs 2/Waitlist (WL) Group; Test type: Superiority; p = 0.042, ANOVA

10. Secondary Outcome: Measure of Pain Inflexibility Pre- and Post-treatment
Description: Pre- and post-treatment pain interference was assessed using the 12-item Psychological Inflexibility in Pain Scale (PIPS). Participants rate their avoidance of activities because of their pain on a Likert scale of 1 (never true) to 7 (always true). Eight of the items are summed to yield a score on the Avoidance subscale, and four of the items are summed for the Fusion subscale. A total score also is obtained by summing all 12 items. We analyzed only the total score in this study, which can range from 12-84, with higher scores indicating more inflexibility (worse).
Time Frame: Baseline and 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1/Acceptance and Commitment Therapy (ACT) Group | 2/Waitlist (WL) Group
Number analyzed (Participants) | 32 | 30
score on a scale
  Baseline | 48.63 (14.8) | 51.53 (14.5)
  8 weeks | 40.10 (13.8) | 49.13 (16.9)

11. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events
Description: Here is the number of participants with serious and non-serious adverse events. A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Baseline, and Week 8, 16, 32, and 40.
Population: Per protocol - "adverse events occurring as a result of treatment for the underlying condition or medical treatment for pain will NOT be recorded or reported on this study." 30/34 were analyzed in the Waitlist group because 2 participants were withdrawn from final analyses due to medical contraindications identified immediately after the post-intervention follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Acceptance and Commitment Therapy (ACT) Group | 2/Waitlist (WL) Group
Number analyzed (Participants) | 32 | 30
Participants
  Baseline | 0 | 0
  Week 8 | 0 | 0
  Week 16 | 0 | 0
  Week 32 | 0 | 0
  Week 40 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline, Week 8, 16, 32, and 40.
Description: Per protocol - "adverse events occurring as a result of treatment for the underlying condition or medical treatment for pain will NOT be recorded or reported on this study."
Arm/Group | 1/Acceptance and Commitment Therapy (ACT) Group | 2/Waitlist (WL) Group
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/34
Other Adverse Events (participants affected / at risk) | 0/32 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/39/NCT02471339/Prot_SAP_000.pdf
  • Informed Consent Form: Assent (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/39/NCT02471339/ICF_001.pdf
  • Informed Consent Form: Standard Consent (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/39/NCT02471339/ICF_002.pdf
  • Informed Consent Form: Screening Consent (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/39/NCT02471339/ICF_003.pdf